CLINICAL TRIAL: NCT06535386
Title: Incidence of Polyuria Associated With Dexmedetomidine During the Intra-operative Period
Brief Title: Polyuria Associated With Dexmedetomidine in Operating Room
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Other Study IDs: HPC
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Polyuria
Keywords: dexmedetomidine; polyuria; anesthesia
MeSH Terms: conditions — Polyuria | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Dexmedetomidine 0.004 MG/ML — Incidence of polyuria during the intraoperative period, associated with dexmedetomidine .

SUMMARY:
Dexmedetomidine is an a2-adrenergic receptor agonist drug, widely used in intensive care for the sedation of patients on mechanical ventilation, as well as in the operating room during invasive procedures and during general anesthesia. It also has anti-inflammatory properties and reduces the need for opioids and benzodiazepines, which leads to a lower incidence of delirium associated with these drugs.

Among the frequent adverse effects associated with the administration of dexmedetomidine we can find bradycardia and hypotension, while some studies carried out in animals have shown that it can increase the diuretic rate.

Polyuria related to pharmacological agonism of a2-adrenergic receptors has been described in vitro and in studies performed in animal models, and is believed to be the result of functional antagonism of arginine vasopressin. Despite its widespread use as a sedative and adjunctive anesthetic, there are very few reports in the literature of dexmedetomidine-related polyuria in humans.

Currently there are no reports in the literature on the incidence of polyuria induced by the intraoperative administration of dexmedetomidine.

DETAILED DESCRIPTION:
This is a prospective, observational study designed to determine the incidence of polyuria, defined as urine output greater than 150 ml/h or 3 ml/kg/h, associated with the administration of dexmedetomidine during the intraoperative period.

The investigators will prospectively and consecutively study all patients scheduled for high complexity surgery under general anesthesia for a period of 4 months.

The diuretic rate will be quantified in ml/hour. A urine sample will be taken two hours after the start of surgery to assess sodium and urinary density, and an arterial blood sample will be taken to determine serum sodium.

Hydration will be recorded in milliliters per hour, detailing the type of solution used.

All data obtained will be captured in a RedCap data collection form.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Scheduled surgery
* Dexmedetomidine in boluses and/or continuous infusion during intra-operative period
* Patients who require arterial line and urinary catheter

Exclusion Criteria:

* Chronic renal disease.
* eGFR < 60 ml/min/1.73m2 for more than 3 months of evolution.
* Emergency or unscheduled surgeries.
* Central nervous system disease at the sellar or suprasellar level.
* Patients receiving diuretics.
* Liver cirrhosis.
* Adrenal gland disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sex and age, over 18-year-old, ASA I - II - III scheduled for high complexity surgery under general anesthesia who receive dexmedetomidine intra-operatively and who require arterial line and urinary catheter, for a period of 4 months.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of polyuria associated with the administration of dexmedetomidine | 3 hours
  Determine the incidence of polyuria defined as urine output greater than 150 ml/h or 3 ml/kg/h associated with the administration of dexmedetomidine during the intraoperative period in patients scheduled for highly complex surgery

SECONDARY OUTCOMES:
determine if the appearance of polyuria is associated with other factors | 3 hours
  Determine if there is any correlation between the appearance of polyuria associated with the administration of dexmedetomidine and age, sex, type of surgery, other anesthetic drugs, and esophageal temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Acosta, MD, Principal Investigator — Hospital Privado de Comunidad

IPD SHARING:
Plan to Share IPD: Undecided